CLINICAL TRIAL: NCT03216291
Title: Home Versus Office Biofeedback Therapy for Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Satish Rao, Professor of Medicine, Division Chief Fellowship Program Director Director, Digestive Health Center, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HomeVOfficeFI
Record Dates: First submitted 2015-10-28; First posted 2017-07-13 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Everyone is masked to the assignment of home or office biofeedback training. Once the subject makes it to their treatment session, then everyone will know which one the subject has been allocated to.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home Biofeedback (Active Comparator): Patients will be given home biofeedback device (InTone) to take home and practice biofeedback exercises at least twice a day for six weeks of therapy. Intervention: Home device biofeedback training.
  Interventions: Device: Home Biofeedback therapy
- Office biofeedback (Active Comparator): Patients with fecal incontinence will receive traditional office biofeedback, once weekly, over six weeks. Intervention: Regular office biofeedback training with assistance of biofeedback person..
  Interventions: Behavioral: biofeedback therapy

INTERVENTIONS:
Behavioral: biofeedback therapy — Biofeedback therapy is a labor-intensive, multi-disciplinary, team approach for the management of patients with anorectal problems. Complete training sessions once a week for 6 weeks in the office.
  Other Names: Training
  Arms: Office biofeedback
Device: Home Biofeedback therapy — Biofeedback therapy is a labor-intensive, multi-disciplinary, team approach for the management of patients with anorectal problems, but instead of an office therapy, the subject will use a biofeedback device to gain strength in their anorectal muscles. This device will be taught how to use in the first session and then the subject will take it home to complete at least 1 session a day for 6 weeks.
  Arms: Home Biofeedback

SUMMARY:
Biofeedback therapy is a labor-intensive, multi-disciplinary, team approach for the management of patients with Fecal Incontinence. It is not easily available to the vast majority of patients in the community with this problem. It is therefore imperative that a more pragmatic therapeutic approach that can be administered easily in the community ought to be developed. However, whether a treatment program that is based on home-training can be just as useful as office-based training has not been evaluated. The purpose of this study is to assess whether having patients train their pelvic floor muscles at home is as effective as in-office biofeedback training.

DETAILED DESCRIPTION:
The specific hypotheses that will be tested are:

1. Home training produces a similar degree of improvement as office biofeedback in

1. overall number of episodes of fecal incontinence
2. normalization of anorectal manometric pressures
3. Overall quality of life and symptom perception on previously validated Fecal Incontinence questionnaires

Thirty patients with fecal incontinence will be recruited for this eight week therapeutic investigation. Fecal Incontinence will be defined as at least 1 episode of solid or liquid stool leakage per week. All patients will provide a detailed history and undergo physical examination, structural (colonoscopy within 10 years) and anorectal manometry. Once eligible for screening, they will sign a consent form and maintain a 2-week prospective stool diary. If the diary confirms Fecal Incontinence and the inclusion criteria are met, they will be enrolled into the study.

After enrollment, patients will be randomized to receive either office-based biofeedback therapy or home-training.

Office-Training: Patients randomized to receive office-based biofeedback therapy will receive an outpatient treatment of neuromuscular pelvic-floor conditioning using biofeedback techniques. In order to improve the pelvic floor muscle coordination and abdominal effort during defecation, patients will be taught pelvic floor and abdominal muscle coordination exercise. Here, the patients are taught to perform kegal-type exercises as well as distend the abdomen by inhaling slowly and then to hold their breath for at least 15 seconds. They are asked to practice this maneuver for 20 minutes, two or three times a day. Patients will be asked to attend the motility laboratory, approximately once every week. Biofeedback therapy will be performed at these clinic office visits by placing a manometry probe that consists of three pressure sensors and a balloon into the anorectum. The pressure sensors are located at 1cm and 2.5 cm from the anal verge and the rectal sensor at 9cm. A 4 cm long latex balloon will be fashioned around the rectal sensor. After probe placement, the patient will remain clothed and seated on a commode in front of a monitor throughout the study.

Anal and pelvic floor muscle training: The goal is to improve the strength coordination and isolation of pelvic floor muscles. Firstly, patients are instructed to isolate the anal sphincter and puborectalis muscles and improve its strength by using modified Kegel exercises in the sitting or lying position with a probe inserted. Visual and verbal feedback techniques are used to reinforce the maneuvers, as they are being performed. The anal and rectal pressure changes displayed on the monitor provides visual feedback to the patient. The verbal feedback is provided by the therapist and consists of either complimenting the patient for performing a correct maneuver or rectifying any errors. The patient is instructed to squeeze and to maintain the squeeze for as long as possible. During the maneuver, the patient observes the monitor and is educated about the changes in anal pressure/EMG activity. For comparison, a normal recording is shown. As the sphincter strength improves, the patient is encouraged to maintain a voluntary contraction for at least 30 seconds. Patients are instructed not to use their abdominal or gluteal muscles to achieve a voluntary squeeze. After a few sessions, the patient is encouraged to perform these maneuvers without visual feedback. The patient is also instructed to perform squeeze exercises at home for at least 20 minutes, two to three times a day, and to perform about 20 squeeze maneuvers per session. Training may be discontinued when patients demonstrate: A reduction in the number of incontinence episodes and improvement in anal squeeze pressure and recto-anal coordination when squeezing. Patients also receive sensory-motor coordination training. The objective here is to achieve a maximum voluntary squeeze in less than 1 second after inflation of a rectal balloon and to control the reflex anal relaxation by consciously contracting the sphincter muscles.

Those randomized to receive home-training will first receive advice regarding standard treatment for fecal incontinence as described previously. Also, they will be asked to attend the motility lab every two weeks to check on the training parameter and recheck the electrical stimulation intensity if it is still appropriate for the training.

During this session, they will be educated regarding the use of the home-trainer device. After general instructions, the investigators will place a reusable, manometry attached with electrical transducer probe into their rectum. Patients will be fitted with Velcro straps that the research team will assist in fitting the patient for. These Velcro straps will allow the probe to stay in place so that the patient will not be required to hold the probe in place throughout the entire training session and thus free up their dominant hand. The probe will be connected to a hand- held pressure sensing device and battery charged monitor with color illuminations to indicate the patient's response.

This is an FDA approved device for use in fecal incontinence. Next, the patient will be asked to lay down on the side of their non-dominant hand, and with their dominant hand they will inflate the manometry probe to a level they consider comfortable, tolerable and "full". If the patient reports this feeling to be tolerable for sustained daily exercise, this volume level will be recorded and maintained for their first two weeks of at home training. Patients will then self-stimulate electrical transducers on the probe to a level they consider tolerable for sustained at-home exercise. This level will also be used for their electrical stimulation throughout their first two weeks of in-home training. At this time the patient is ready to begin their first training session. The device will provide voice-guided instructions for the patients self-directed biofeedback exercise, as well as visual and audio feedback during these pelvic floor muscle toning exercises. Thus, by observing the number of lights that are activated, the patient receives instant feedback about their performance. Initially, the electrical simulations will be set at the highest initial comfortable level for most individuals. Thereafter, at subsequent office visits, appropriate adjustments will be made and suitable targets designed for each patient to achieve the desired goal of pelvic floor strengthening.

The patient will be instructed by the InTone device's training paradigm, at least twice a day and practice a minimum of 20 minutes of 10 second sustained squeezing then follow by 5 minutes of rectal electrical stimulation with the device.

After each use, the probe can be rinsed with soap and water and reused. The training device is battery powered and can be recharged. Once charged the power lasts for at least 30 days and should facilitate the use of this device between office follow-up sessions.

Patient compliance will be automatically monitored and stored in the device recorder. After two weeks of home-training, the patients will return for a follow up assessment and exercise compliance will be reviewed. Based on their progress, newer targets will be set by adjusting the electrical stimulation levels of the training device. During this visit, any other problems or issues will also be addressed. Four weeks later they will be asked to return again and during this visit a repeat anorectal manometry assessment will be performed and patients will complete post-treatment questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* recurrent episodes of fecal incontinence for six months
* no mucosal disease
* on a two week stool diary patient will report at least one episode of incontinence a week

Exclusion Criteria:

* severe diarrhea
* on opioids, tricyclics (except on stable doses > 3months)
* active depression
* comorbid illnesses, severe cardiac disease, chronic renal failure or previous gastrointestinal surgery except cholecystectomy and appendectomy
* neurologic diseases (e.g. head injury, epilepsy, multiple sclerosis, strokes, spinal cord injury)
* impaired cognizance (mini mental score of < 15) and/or legally blind
* metal implants, pacemakers
* previous pelvic surgery, bladder repair, radical hysterectomy
* ulcerative and Crohn's colitis
* rectal prolapse, anal fissure, anal surgery or inflamed hemorrhoids
* pregnant women or nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Number of episodes of fecal incontinence | six weeks
  Assess the change in the No of FI episodes between baseline week and end of study week and compare between the two treatment groups. Responder is defined as a patient with greater than 50% reduction in FI episodes after treatment when compared to baseline. Responder rates will compared between the two treatment groups.

SECONDARY OUTCOMES:
Overall quality of life and symptom perception on previously validated Fecal Incontinence questionnaires | six weeks
  Assess the change in 4 quality of life domains between baseline SF-11 survey and survey done at the end of treatment and compare between the 2 treatment groups
Anal sphincter pressure and rectal sensation | six weeks
  Assess the changes in anal resting and squeeze sphincter pressures (mmHg) and sensory data between baseline anorectal manometry study and study done at the end of treatment and compare between the 2 treatment groups.
FI severity, quality of life and bowel symptoms | Six weeks
  The FI severity and quality of life and bowel symptoms will be assessed using ICIQ-B, FISS, FISI questionnaires (numerical mean scores for individual questions or groups of questions) and compared between two groups.
Treatment compliance with home biofeedback | Six weeks
  The treatment compliance will be assessed by examining daily logs of computer which includes the duration and completion of each home biofeedback session.

CONTACTS AND LOCATIONS:
Overall Officials: Satish Rao, MD, PhD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No